CLINICAL TRIAL: NCT03070080
Title: Restrictive Versus Conservative Fluid Therapy in Colorectal Surgery: Hemodynamics and Kidney Function Outcomes
Brief Title: Restrictive Versus Conservative Fluid Therapy in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdel-Baky Abdel-Rahman, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23140000178
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2017-03

CONDITIONS: Fluid Therapy
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- restrictive group (Active Comparator): restrictive fluid strategy, 6 ml/kg/hour of lactated Ringer, during intraoperative period
  Interventions: Procedure: restrictive fluid strategy
- conservative group (Active Comparator): conservative fluid strategy, 12 ml/kg/hour of lactated Ringer, during intraoperative period
  Interventions: Procedure: conservative fluid strategy

INTERVENTIONS:
Procedure: restrictive fluid strategy — restrictive lactated ringers as intraoperative fluid therapy in a dose of 6ml/kg/hour
  Other Names: fluid therapy
  Arms: restrictive group
Procedure: conservative fluid strategy — conservative lactated ringers as intraoperative fluid therapy in a dose of 12ml/kg/hour
  Other Names: conservative fluid therapy
  Arms: conservative group

SUMMARY:
Fluid administration during and after surgery is an essential part of postoperative care to maintain the patients' fluid and biochemical balance. Abdominal surgical procedures are associated with dehydration from preoperative fasting, bowel preparation, and intra- and postoperative fluid and electrolyte loss. So, perioperative fluid management has been a topic of much debate over years and has intensified especially over the past several years.

DETAILED DESCRIPTION:
The controversies include the type of fluid, the timing of administration and the volume administrated. Following much discussion and ongoing controversy on colloids versus crystalloids and the ideal composition of the various intravenous solutions, the main focus more recently has been on the volume of fluids.

Fluid therapy strategies have been developed and implemented in clinical practice over several decades. The data suggest that aggressive or liberal intraoperative fluid resuscitation is harmful during open abdominal operation, whereas a restrictive fluid protocol has better outcomes, including fewer postoperative complications and a shorter discharge time.

However, a restrictive fluid regimen has several limitations. Overly restricted or inadequate fluid administration may lead to insufficient intravascular volume, tissue hypoperfusion, cellular oxygenation impairment and potential organ dysfunction, prolonged recovery of bowel function, and impair tissue oxygenation, which might ultimately impair wound healing including healing of anastomosis.

Recently, the pleth-variability index (PVI) derived from respiratory variations in peripheral perfusion index (PI) has been suggested to be an effective dynamic indicator of fluid responsiveness. Different from other invasive dynamic indices, PVI provides clinicians with a numerical value obtained non-invasively. PVI is calculated as [(PI max - PI min)/PI max] X 100, where PI max and PI min represent the maximal and the minimal value, respectively, of the plethysmographic perfusion index (PI) over one respiratory cycle. PI is the ratio between pulsatile and non-pulsatile infrared light absorption from the pulse oximeter, and it is physiologically equivalent to the amplitude of the plethysmographic waveform. A PVI value of >13% before volume expansion discriminated between fluid responders and non responders with 81% sensitivity and 100% specificity.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients scheduled for colorectal surgery
2. American Society of Anesthesiologists grade I-II.

Exclusion criteria:

1. patient refusal.
2. psychiatric disorders.
3. pregnancy and lactation.
4. preexisting neurological dysfunction ( history of cerebrovascular stroke CVS)
5. Allergy to any protocol medication.
6. metastatic cancer.
7. Inflammatory bowel disease.
8. Coronary artery disease with impaired cardiac function.
9. Diabetes mellitus.
10. Renal insufficiency (serum creatinine level more than 180 μmol/l).
11. unexpected intraoperative findings (small bowel obstruction, inoperable).
12. accidental massive intraoperative haemorrhage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Neutrophil Gelatinase-associated Lipocalin (NGAL) | 24 hours postoperative
  NGAL is a renal biomarker for acute kidney injury

SECONDARY OUTCOMES:
mean arterial blood pressure | intraoperative
  non invasive measurement of mean arterial blood pressure
heart rate | intraoperative
  measurement of heart rate from pulse oximetry
pleth-variability index | intraoperative
  derived from respiratory variations in peripheral perfusion index.
incidence of bradycardia | intraoperative
  bradycardia defined as heart rate less than 50 beat per minute
incidence of hypotension | intraoperative
  hypotension defined as systolic blood pressure less than 40% of baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Abdel-Rahman, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut Iniversity hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided